CLINICAL TRIAL: NCT03644264
Title: An Open-label, Randomised, Active-controlled, Parallel Group, Multicentre, Phase 3 Study to Investigate the Safety and Efficacy of PA21 and Sevelamer Carbonate (Renvela®) in Chinese CKD Patients With Hyperphosphataemia
Brief Title: PA21 Safety and Efficacy in Adult Chinese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor Fresenius Medical Care Renal Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA-CL-CHINA-01
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis; Hyperphosphatemia
Keywords: Chronic Kidney Disease; Hyperphosphatemia; Dialysis
MeSH Terms: conditions — Hyperphosphatemia; Renal Insufficiency, Chronic | interventions — sucroferric oxyhydroxide; Sevelamer

STUDY DESIGN:
Intervention Model Description: Open-label, Randomised, Active-controlled, Parallel Group, Multicentre,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PA21 tablets containing 500 mg of iron (Experimental): PA21 chewable tablets standardised to contain 500 mg of iron. PA21 500 mg (iron) chewable tablet contains approximately 2.5 g PA21 drug substance (sucroferric oxyhydroxide). Starting dose will be 1,500 mg/day (3 tablets/day (1 tablet per meal)). Dose increases or decreases of 500 mg/day (1 tablet/day) are permitted. The maximum dose of PA21 will be 3,000 mg/day (6 x 500 mg tablets/day) and the minimum dose will be 1,000 mg/day (2 x 500 mg tablets/day).
  Interventions: Drug: PA21
- Sevelamer carbonate: Renvela® tablets (Active Comparator): Starting dose will be 2.4 g/day (3 tablets/day). Dose increases or decreases of 2.4 g/day (3 tablets/day (1 tablet per meal)) The maximum dose of sevelamer carbonate will be 14.4 g/day (18 tablets/day) and the minimum dose will be 2.4 g/day (3 tablets/day).
  Interventions: Drug: sevelamer carbonate

INTERVENTIONS:
Drug: PA21 — sucroferric oxyhydroxide is a mixture of polynuclear iron(III)-oxyhydroxide (about 33% m/m), sucrose (about 30% m/m), and starches (about 28% m/m) and contains ≤10% m/m water.
  Other Names: sucroferric oxyhydroxide; Velphoro®
  Arms: PA21 tablets containing 500 mg of iron
Drug: sevelamer carbonate — sevelamer carbonate tablets containing 800 mg of sevelamer carbonate.
  Other Names: Renvela®
  Arms: Sevelamer carbonate: Renvela® tablets

SUMMARY:
This study evaluates the efficacy of PA21 in comparison with sevelamer carbonate (Renvela®) in lowering and maintaining serum phosphorus in adult Chinese subjects with CKD on dialysis after 12 weeks of treatment.

DETAILED DESCRIPTION:
Primary Objective is to evaluate the efficacy of PA21 in comparison with sevelamer carbonate (Renvela®) in lowering and maintaining serum phosphorus in adult Chinese subjects with CKD on dialysis after 12 weeks of treatment. In addition , secondary objectives include evaluating the efficacy of PA21 and sevelamer carbonate over time as the percentage of subjects with serum phosphorus within the target range of 1.13 to 1.78 mmol/l (3.5 to 5.5 mg/dl) and to compare the safety and tolerability of PA21 versus sevelamer carbonate (Renvela®).

In total, 286 patients (143 patients to PA21 treatment and 143 patients to sevelamer carbonate treatment) will be randomised with a screening period: up to 4 weeks and a washout period of up to 3 weeks. Treatment period (total duration 12 weeks) will include a dose titration period and a maintenance period of an open-label, active-controlled comparison of PA21 versus sevelamer carbonate for 4 weeks. The primary efficacy assessment will be a non-inferiority assessment of the 2 groups of subjects at Week 12 in terms of serum phosphate lowering capability. There will be a follow-up period of 30 days after last dosing.

The investigational treatments will be a PA21 dose group of PA21 chewable tablets standardised to contain 500 mg of iron. PA21 contains approximately 20% m/m of elemental iron. All doses of PA21 are expressed in mg of iron. The Starting dose will be 1,500 mg/day (3 tablets/day (1 tablet per meal)). Dose increases or decreases of 500 mg/day (1 tablet/day) are permitted , provided a subject has been receiving that dose for a minimum of 2 weeks and for safety or tolerability reasons at any time. The maximum dose of PA21 will be 3,000 mg/day (6 x 500 mg tablets/day) and the minimum dose will be 1,000 mg/day (2 x 500 mg tablets/day). The active control is sevelamer carbonate, Renvela®, tablets, containing 800 mg of sevelamer carbonate. The starting dose will be 2.4 g/day (3 tablets/day). Dose increases or decreases of 2.4 g/day (3 tablets/day (1 tablet per meal)) are permitted, provided a subject has been receiving that dose for a minimum of 2 weeks, and for safety or tolerability reasons at any time. The maximum dose of sevelamer carbonate will be 14.4 g/day (18 tablets/day) and the minimum dose will be 2.4 g/day (3 tablets/day).

ELIGIBILITY:
Inclusion Criteria:

1. Chinese subjects receiving either maintenance haemodialysis (HD) or peritoneal dialysis (PD) for at least 12 weeks prior to screening. No home HD or nocturnal HD (overnight stay at site) will be allowed
2. Subjects with a history of hyperphosphataemia (HP).
3. Subjects with serum phosphorus levels >5.5 mg/dl (>1.78 mmol/l) at screening or during the washout period.
4. Male and female adult subjects (aged ≥18 years at time of consent).
5. Subjects with the ability to understand the requirements of the study and abide by the study restrictions, and who agree to return for the required assessments (in the Investigator's opinion).
6. Subject (or legally acceptable representative) has provided the appropriate written informed consent. Subject must provide written informed consent before any study-specific procedures are performed including screening procedures.

Exclusion Criteria:

1. Subjects with intact parathyroid hormone (iPTH) levels >800 ng/l (>800 pg/ml or 88 pmol/l) at screening. Subjects with iPTH >600 ng/l (>600 pg/ml or 66 pmol/l) at screening must be considered stable (in the Investigator's opinion).
2. Subjects with planned or expected parathyroidectomy within the next 6 months (in the Investigator's opinion).
3. Subjects on peritoneal dialysis (PD) with a history of peritonitis in the last 3 months or ≥3 episodes in the last 12 months.
4. Subjects with serum total calcium >10.5 mg/dl (>2.6 mmol/l) or <7.6 mg/dl (1.9 mmol/l) at screening.
5. Subjects with:

   * Any history of major gastrointestinal (GI) surgery likely to influence the outcome of treatment with PBs
   * Clinically significant, active GI disorders (e.g., active peptic ulcer, Crohn's disease, colitis ulcerative, irritable bowel syndrome, intestinal motility disorder (symptomatic gastroparesis (during treatment or untreated), intestinal obstruction, moderate/severe constipation (including persistent symptoms with regular use of laxatives or enemas and limitations in activities of daily living), intestinal pseudo-obstruction, megacolon, mechanical obstruction)) or any GI disorders under medical treatment.
   * Clinically significant, active hepatic disorders or any hepatic disorder under medical treatment
6. Subjects currently with (in the Investigator's opinion):

   * Swallowing difficulties/dysphagia
   * Estimated life expectancy of less than 12 months
   * Anticipated renal transplantation during study participation
7. Subjects with known seropositivity to human immunodeficiency virus or positive HIV test at screening.
8. Subjects with active/current fulminant hepatitis B infections and/or hepatitis C virus ribonucleic acid positivity at screening.
9. Subjects with a history of haemochromatosis or other iron accumulation disorders that might lead to iron overload.
10. Subjects with serum ferritin >800 mcg/l (1,797.6 pmol/l) or transferrin saturation (TSAT) >50% at screening.
11. Subjects with raised alanine aminotransferase or aspartate aminotransferase >3 times the upper limit of the normal range at screening.
12. Subject is taking any prohibited medication(s) which cannot be stopped at least one week before study treatment start. Prohibited medications include: oral calcium supplements, any drugs/agents having a phosphate binding action that contain aluminium, magnesium or calcium (apart from hyperkalaemia drugs), phosphate binders in addition to sevelamer carbonate), nicotinamide, oral iron products, oral vitamins containing iron and other oral iron containing supplements (See Section 7.7).
13. Subject has known hypersensitivity and/or intolerance to any of the study products to be administered.
14. Subject has previously been randomised into this study.
15. Subject is currently enrolled in or has completed any other investigational device or drug study <30 days prior to screening, or is receiving other investigational agent(s).
16. Subjects who are pregnant (e.g., positive human chorionic gonadotropin test) or breastfeeding.
17. Subjects of childbearing potential, not using adequate contraceptive precautions must agree to use a highly effective method of birth control during the study and for 1 month after the last dose of study medication.
18. Subject has a history of drug or alcohol abuse within 2 years prior to screening.
19. Subject has a significant medical conditions or anticipated need for major surgery during the study, which (in the Investigator's opinion), may be associated with increased risk to the subject, or may interfere with study assessments or outcomes, or the ability to provide informed consent or comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Serum phosphorus (mmol/l ) | baseline and 12 weeks
  Change from baseline in serum phosphorus levels at Week 12: comparison between PA21 group and sevelamer carbonate group.

SECONDARY OUTCOMES:
Serum phosphorus (mmol/l ) | baseline, weeks 1, 2, 4, 6, 8, 12
  Serum phosphorus levels at each time point and change from baseline (BL)
Serum phosphorus (mmol/l) | baseline, weeks 1, 2, 4, 6, 8, 12
  % of subjects with serum phosphorus within 1.13 to 1.78 mmol/l
Adverse events (AEs) | baseline, weeks 1, 2, 4, 6, 8, 12
  Frequency of AEs determined by seriousness, severity and relatedness to study drugs
Diarrhoea. | baseline, weeks 1, 2, 4, 6, 8, 12
  Frequency of AE of special interest - diarrhoea.
Withdrawals due to AEs | baseline, weeks 1, 2, 4, 6, 8, 12
  Percentage of withdrawals due to AEs
Serum calcium (mmol/l) | baseline, weeks 1, 2, 4, 6, 8, 12
  Serum total calcium levels at each time point and change from baseline
Hypercalcemia (mmol/l) | baseline, weeks 1, 2, 4, 6, 8, 12
  Percentage of subjects that develop at least 1 episode of sustained hypercalcaemia (>10.0 mg/dl; >2.5 mmol/l) during study participation
Serum iPTH (pg/ml) | baseline, weeks 8, 12
  Serum iPTH levels at specified time points and change from baseline
Serum iron (mcg/dl) | baseline, weeks 4, 8, 12
  Serum iPTH levels at specified time points and change from baseline
Serum ferritin (mcg/l) | baseline, weeks 4, 8, 12
  Serum ferritin levels at specified time points and change from baseline
Serum transferrin (mcg/dl) | baseline, weeks 4, 8, 12
  Serum transferrin measured at specified timepoints
Transferrin saturation (TSAT) (%) | baseline, weeks 4, 8, 12
  TSAT measured at specified timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Hou Fanfan, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Southern Medical University Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Liu J, Zuo L, Walpen S, Bernard L, Marty M, Enoiu M. Efficacy and Safety of Sucroferric Oxyhydroxide Compared with Sevelamer Carbonate in Chinese Dialysis Patients with Hyperphosphataemia: A Randomised, Open-Label, Multicentre, 12-Week Phase III Study. Nephron. 2024;148(1):22-33. doi: 10.1159/000531869. Epub 2023 Jul 20. PMID 37473746